CLINICAL TRIAL: NCT06283615
Title: Effect of Vitamin D Supplementation on Skeletal Muscle Function and Quality of Life in Patients With Chronic Intestinal Failure/Insufficiency: A Randomised Clinical Trial
Brief Title: Effect of Vitamin D on Skeletal Muscle Function and Qol in Patients With Chronic Intestinal Failure/Insufficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Wang Xinying, Prof, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-01-01
Record Dates: First submitted 2024-01-18; First posted 2024-02-28 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Intestinal Failure
Keywords: Vitamin D; Quality of life; Muscle function; Chronic intestinal failure
MeSH Terms: conditions — Intestinal Failure | interventions — Vitamin D; Ergocalciferols

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin D (Experimental): Experimental group: In addition to conventional treatment, additional intramuscular injection of vitamin D2 was given once every two weeks, each dose of 600,000 units, and the treatment lasted for 12 weeks.
  Interventions: Drug: Vitamin D
- Control (No Intervention): Control group: received appearance-matched placebo plus standard care, no additional vitamin D intervention therapy.

INTERVENTIONS:
Drug: Vitamin D — Vitamin D2 injection
  Other Names: Vitamin D2
  Arms: Vitamin D

SUMMARY:
Eligible patients were randomized into two groups: Vitamin D group and Control group. Control group: received placebo plus standard care, no additional vitamin D intervention therapy. Vitamin D group: In addition to the standard care, additional intramuscular injection of vitamin D2 was given once every two weeks, each dose of 600,000 units, and the treatment lasted for 12 weeks.

The primary and secondary outcomes will be collected.

DETAILED DESCRIPTION:
Eligible patients with chronic intestinal failure/insufficiency were randomly assigned to one of two groups, Vitamin D group and Control group. Control group: received placebo plus standard care, no additional vitamin D intervention therapy. Vitamin D group: In addition to the conventional treatment, additional intramuscular injection of vitamin D2 was given once every two weeks, each dose of 600,000 units, and the treatment lasted for 12 weeks.

The primary and secondary outcomes will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent was obtained from patients or their legal representatives for participation in this study
2. Patients 18 years of age or older, under 70 years of age, chronic intestinal failure/insufficiency
3. Serum 25(OH)D level < 30.0 ng/ml
4. Vital signs are stable

Exclusion Criteria:

1. Those who did not meet the inclusion criteria, or who were deemed unfit by their physician to participate in this study
2. Primary hypothyroidism or parathyroidism
3. Patients suffering from allergic diseases, are allergic, have a history of drug sensitivity similar to the structure of the study drug
4. Patients with primary diabetes
5. Patients with mental illness, inability to cooperate or consciousness disorders
6. Patients with contraindications of experimental drugs
7. Patients with a suspected or confirmed history of substance abuse
8. Immune deficiency, use of immunosuppressants and hormones
9. Pregnant and lactating women
10. Have taken any vitamin D supplements in the last 6 months
11. Have taken any medication in the last 6 months that affects vitamin D metabolism (e.g., phenytoin, phenobarbital, rifampicin)
12. Patients who participated in a drug trial (including the drug in the trial) within 3 months before the trial
13. Sponsors or investigators directly involved in the trial or their family members
14. The researcher believes that there is any reason not to be accepted

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2024-03-12 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Quality of life score | up to 12 weeks
  Quality of life was assessed using the SF-36 score from the date of randomization until the end of the 12-week intervention weeks. SF-36 consists of eight dimensions, each of which is measured on a scale of 0-100, with higher scores indicating a better quality of life.
Muscle function status | up to 12 weeks
  Including hand grip strength(kg); Appendicular skeletal muscle mass index (ASMI) = limb muscle mass (kg)/height (m)2；6 meters walking speed(m/s)

SECONDARY OUTCOMES:
Serum vitamin D levels | up to 12 weeks
  Serum 25 hydroxyvitamin D levels
Hepatic and renal function | up to 12 weeks
  Liver function includes the following indicators: Alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin (TBil), direct and indirect bilirubin, γ-glutamyltranspeptidase (γ-GT) and alkaline phosphatase (ALP). Kidney function includes the following indicators: serum creatinine and blood urea nitrogen.
Bone mineral density | up to 12 weeks
  Bone mineral density by DXA
Thyroid and parathyroid-related hormones | up to 12 weeks
  Including surum total triiodothyroxine, total tetraiodothyroxine, free triiodothyronine, free tetraiodothyroxine, thyroid stimulating hormone, parathyroid hormone and calcitonin.
Nutritional status indicators | up to 12 weeks
  Including body weight (kg), serum albumin (g/L) and prealbumin (mg/L) levels.
Number of participants with treatment-related adverse events | up to 12 weeks
  Occurrence of hypercalcemia and hyperphosphatemia during intervention and follow-up. The blood calcium concentration > 2.75 mmol/L is called hypercalcemia. Normal human blood phosphorus concentration is relatively stable (normal reference value 0.87~1.45mmol/ L), when the determination result is greater than the normal reference value of 1.45mmol/ L, it can be diagnosed as hyperphosphatemia.
  Occurrences of kidney stones during intervention and follow-up. Kidney stones are examined by ultrasound.
  Incidence of fall-related fractures during intervention and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Xinying Wang, MD, Principal Investigator — Jinling Hospital, China
Locations (1):
- Xinying Wang, Nanning, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pironi L, Corcos O, Forbes A, Holst M, Joly F, Jonkers C, Klek S, Lal S, Blaser AR, Rollins KE, Sasdelli AS, Shaffer J, Van Gossum A, Wanten G, Zanfi C, Lobo DN; ESPEN Acute and Chronic Intestinal Failure Special Interest Groups. Intestinal failure in adults: Recommendations from the ESPEN expert groups. Clin Nutr. 2018 Dec;37(6 Pt A):1798-1809. doi: 10.1016/j.clnu.2018.07.036. Epub 2018 Aug 18. PMID 30172658
- [Background] Khan FA, Fisher JG, Bairdain S, Sparks EA, Zurakowski D, Modi BP, Duggan C, Jaksic T. Metabolic bone disease in pediatric intestinal failure patients: prevalence and risk factors. J Pediatr Surg. 2015 Jan;50(1):136-9. doi: 10.1016/j.jpedsurg.2014.10.010. Epub 2014 Oct 17. PMID 25598110
- [Background] Yang CF, Duro D, Zurakowski D, Lee M, Jaksic T, Duggan C. High prevalence of multiple micronutrient deficiencies in children with intestinal failure: a longitudinal study. J Pediatr. 2011 Jul;159(1):39-44.e1. doi: 10.1016/j.jpeds.2010.12.049. Epub 2011 Feb 16. PMID 21324480
- [Background] Reid IR, Bolland MJ, Grey A. Effects of vitamin D supplements on bone mineral density: a systematic review and meta-analysis. Lancet. 2014 Jan 11;383(9912):146-55. doi: 10.1016/S0140-6736(13)61647-5. Epub 2013 Oct 11. PMID 24119980
- [Background] Holick MF. Sunlight and vitamin D for bone health and prevention of autoimmune diseases, cancers, and cardiovascular disease. Am J Clin Nutr. 2004 Dec;80(6 Suppl):1678S-88S. doi: 10.1093/ajcn/80.6.1678S. PMID 15585788
- [Background] Lepus CA, Samela K, Emerick KM, Mokha JS. Vitamin D status in children with intestinal failure who have achieved enteral autonomy. Nutr Clin Pract. 2021 Dec;36(6):1284-1289. doi: 10.1002/ncp.10685. Epub 2021 Jun 23. PMID 34161622
- [Background] Wozniak LJ, Bechtold HM, Reyen LE, Hall TR, Vargas JH. Vitamin D deficiency in children with intestinal failure receiving home parenteral nutrition. JPEN J Parenter Enteral Nutr. 2015 May;39(4):471-5. doi: 10.1177/0148607114527135. Epub 2014 Mar 14. PMID 24633203
- [Background] Allan PJ, Lal S. Metabolic bone diseases in intestinal failure. J Hum Nutr Diet. 2020 Jun;33(3):423-430. doi: 10.1111/jhn.12726. Epub 2019 Dec 11. PMID 31823437
- [Background] Diamanti A, Capriati T, Cardile S, Benedetti S, Francalanci P, Elia D. Fat-soluble vitamin deficiency in children with intestinal failure receiving home parenteral nutrition. J Pediatr Gastroenterol Nutr. 2014 Nov;59(5):e46. doi: 10.1097/MPG.0000000000000508. No abstract available. PMID 25347160